CLINICAL TRIAL: NCT07174609
Title: A Pilot Study of Scrambler Therapy for Painful Chronic Pancreatitis
Brief Title: Scrambler Therapy in Chronic Pancreatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The National Pancreas Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00469056
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Pancreatitis; Chronic Pancreatitis
Keywords: chronic pain; Abdominal pain; chronic pancreatitis; Scrambler Therapy; Electrocutaneous analgesia
MeSH Terms: conditions — Chronic Pain; Pancreatitis; Pancreatitis, Chronic; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: This is a single-arm feasibility study using a Single Group Assignment design. All participants with chronic pancreatitis and refractory abdominal pain will receive Scrambler Therapy, consisting of 5-10 daily treatment sessions lasting 30-40 minutes. There is no randomization or control arm. Outcomes will include feasibility measures (enrollment, adherence, and retention), as well as changes in pain severity, opioid use, and patient-reported quality of life over 3 months of follow-up. The purpose is to generate preliminary safety and effectiveness data to support future controlled trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Scrambler Therapy for Chronic Pancreatitis Pain (Experimental): Adults with chronic pancreatitis and refractory abdominal pain will receive Scrambler therapy. Scrambler Therapy is a non-invasive neuromodulation treatment designed to relieve chronic pain by transmitting "non-pain" electrical signals through the skin to the nervous system. The device generates 16 variable waveforms that mimic natural nerve impulses, creating patient-specific cutaneous electrostimulation. These signals are carried by afferent C-fibers and interpreted by the central nervous system as non-painful, thereby modulating pain perception rather than blocking it.
  Interventions: Device: Scrambler Therapy

INTERVENTIONS:
Device: Scrambler Therapy — Adults with chronic pancreatitis and refractory abdominal pain will receive Scrambler Therapy, a non-invasive neuromodulation device. Electrodes are placed near the painful area to deliver "non-pain" signals aimed at reducing pain perception. Participants will complete 5-10 daily treatment sessions, each lasting 30-40 minutes, with pain ratings collected before and after sessions and follow-up assessments over 3 months.

SUMMARY:
The investigators will enroll adults with chronic pancreatitis who have persistent abdominal pain not relieved by standard treatments. This study will test the feasibility and effectiveness of Scrambler Therapy, a non-invasive FDA-cleared device that delivers "non-pain" electrical signals through the skin to retrain the brain's pain perception. Participants will undergo 5-10 treatment sessions and be followed for 3 months with standardized pain scores and quality-of-life assessments. The goal is to generate pilot data to support larger studies of Scrambler Therapy as a novel option for pancreatic pain.

DETAILED DESCRIPTION:
This is a single-arm, observational pilot study to test whether Scrambler Therapy (ST) is a feasible and effective treatment for refractory abdominal pain in chronic pancreatitis. Approximately 40 adults with Chronic Pancreatitis (CP) will be enrolled through outpatient clinics and inpatient consults. Eligible participants are those who continue to experience significant pain despite medical and/or endoscopic or surgical management.

After informed consent, participants will undergo 5-10 daily Scrambler Therapy sessions lasting 30-40 minutes each. Electrodes will be placed on skin areas near, but not directly over, the sites of pain. Treatment intensity will be adjusted until patients perceive a tolerable, tingling "non-pain" sensation. Pain ratings (0-10 visual analogue scale, VAS) will be collected before and after each session.

Participants will be followed for 3 months, with weekly pain ratings collected via text, phone, or email, and standardized questionnaires at 3 months. Secondary outcomes include opioid use, 30% and 50% pain reduction, and patient-reported outcomes (PROMIS tools and Patient Global Impression of Change). Safety will be monitored by recording any adverse events, with particular attention to mild skin irritation at electrode sites.

The primary goal is to determine the feasibility of enrolling and retaining patients and their willingness to complete treatment and follow-up. If Scrambler Therapy shows promise, these data will support the design of larger controlled trials aimed at improving pain management for patients with chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosis of chronic pancreatitis with refractory abdominal pain
* Able to provide written informed consent in English
* Sufficient English language ability to complete study questionnaires
* Reliable and regular access to a phone for follow-up

Exclusion Criteria:

* Unable or unwilling to provide written consent
* History or presence of a significant medical or psychiatric condition that would interfere with study participation
* Pregnant or lactating women
* Coronary stents or implanted metallic/electrical devices (pacemaker, defibrillator, aneurysm clips)
* History of epilepsy, traumatic brain injury, or myocardial infarction within the past 6 months
* Skin conditions preventing electrode placement (e.g., open wounds)
* Any condition that, in the investigator's opinion, places the participant at increased risk or prevents full compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by enrollment rate | During recruitment ( expected 24 months)
  Number of eligible patients who consent and enroll divided by the total number of eligible patients approached.
Feasibility as assessed by treatment adherence | During treatment period (up to 2 weeks)
  Number of participants who complete a minimum of 5 Scrambler Therapy sessions out of the planned 5-10, or who discontinue earlier due to achieving adequate pain relief.
Feasibility as assessed by treatment adherence rate | During treatment period (average 5-10 days, up to 2 weeks)
  Proportion of participants who complete a minimum of 5 Scrambler Therapy sessions out of the planned 5-10, or who discontinue earlier due to achieving adequate pain relief.
Feasibility as assessed by retention | Baseline through 3 months post-treatment
  Proportion of enrolled participants who complete the 3-month follow-up assessments, including pain ratings.

SECONDARY OUTCOMES:
Change in Pain Intensity (VAS) | Baseline, 1 month, and 3 months after treatment
  Change in abdominal pain severity measured by Visual Analogue Scale (VAS, 0-10).Rating Scale (NRS, 0 = no pain, 10 = worst imaginable pain).
Percentage of Patients with ≥30% Pain Reduction | Baseline , 1 months and 3 months post-treatment
  Percentage of participants achieving at least a 30% reduction in VAS pain score compared with baseline.
Percentage of Patients with ≥50% Pain Reduction | Baseline, 1 month and 3 months post-treatment
  Percentage of participants achieving at least a 50% reduction in VAS pain score compared with baseline.
Opioid use | Baseline, 1 month and 3 months post-treatment
  Number of patients using prescription opioids for pain control at time of assessment
Daily opioid dose( morphine milligram equivalents,MME) | Baseline, 1 month and 3 months post-treatment
  Change in mean daily prescription opioid dose reported by participants, converted to morphine milligram equivalents.
Patient Global Impression of Change (PGIC) | 1 month, 3 months
  PGIC is a 7-point Likert scale (1 = very much improved, 7 = very much worse).
Change from baseline on the Patient Reported Outcomes Measurement Information System (PROMIS) Global Health Scale. | Baseline, 1 month, and 3 months after treatment
  Change from baseline in PROMIS Global Health, which provides physical and mental health scores (range 7-35; higher = better health).
Change from baseline on the Hospital Anxiety and Depression Scale (HADS) | Baseline, 1 month, and 3 months post-treatment
  The HADS is a validated self-reported tool that screens for symptoms of anxiety and depression. Possible scores range from 0 to 21 (higher scores reflect more severe symptoms of anxiety or depression).
Change from baseline on the Modified Brief Pain Inventory Short Form | Baseline, 1 month and 3 months
  Change from baseline in mBPI-SF. Pain severity score range 0-40; pain interference score range 0-70. Higher = worse pain or more interference.
Change from baseline on the European Organization for the Research and Treatment of Cancer Quality(EORTC) of Life Questionnaire (QLQ) Core 30 (C30) | Baseline, 1 month and 3 months
  Change from baseline in European Organization for Research and Treatment of Cancer QLQ-C30 (0-100). Higher = better on global/functioning scales; higher = worse on symptom scales.
Change from baseline on the Comprehensive Pain Assessment Tool for Pancreatitis Short Form (COMPAT-SF) | Baseline, 1 month and 3 months
  Change from baseline in COMPAT-SF. The COMPAT-SF is a validated self-reported tool specifically designed for patients with pancreatic disease. Scores for pain severity (average, worst, and least) range from 0 to 10 (higher corresponds to more pain); scores for pain triggers (including food, exercise, and thermal changes) are scored on a scale from never to always (never, rarely, sometimes, very often, always); scores for pain symptom characteristics (cramping, shooting, stabbing) are scored on a scale from 0 (none) to 10 (worst possible). The total score is a weighted score derived from individual dimension scores which are then normalized to a 0-100 scale.

OTHER OUTCOMES:
Adverse events - Frequency | During treatment ( up to 2 weeks)
  Frequency of treatment-related adverse events, including skin irritation or discomfort at electrode sites.

CONTACTS AND LOCATIONS:
Overall Officials: Mahya Faghih, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Green Spring Station, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No